CLINICAL TRIAL: NCT02735369
Title: A Phase II, Randomized, Placebo-Controlled, Study Assessing Efficacy and Safety of OC-10X Ophthalmic Suspension in the Treatment of Proliferative Diabetic Retinopathy
Brief Title: A Study Assessing Efficacy and Safety of OC-10X in the Treatment of PDR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: OcuCure Therapeutics, Inc. (Industry)
Collaborators: Semler Research Center Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC10X-CT-BD2 PDR
Record Dates: First submitted 2016-01-19; First posted 2016-04-12 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Proliferative Diabetic Retinopathy (PDR)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo Comparator
- 2% OC-10X (Experimental): 2% OC-10X
  Interventions: Drug: 2% OC-10X

INTERVENTIONS:
Drug: 2% OC-10X — 2% OC-10X
  Other Names: 2-Biphenyl-4-yl-2,3-dihydro-(1H)-quinazolin-4-one
  Arms: 2% OC-10X
Drug: Placebo Comparator — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The present study is intended to evaluate the efficacy and safety of topical OC-10X Ophthalmic Suspension in patients diagnosed with proliferative diabetic retinopathy (level 61, 65, 71, or 75). OcuCure Therapeutics, Inc. (Roanoke, VA) has developed a lead compound, known as OC-10X, which is a selective tubulin inhibitor under development for the treatment of Proliferative Diabetic Retinopathy (PDR) and Age-related Macular Degeneration (AMD). When administered as a topical eye drop, OC-10X has both anti-angiogenic (inhibition) and angiolytic (regression) properties in animal models of choroidal neovascularization (CNV). Unlike other therapies, OC-10X provides the efficacy of a vascular targeting agent without the traditional toxicity and works downstream independently of growth factors. As demonstrated by OcuCure's preclinical data, tubulin inhibition, using OC-10X, may be a promising new approach to the treatment of PDR and AMD. Like AMD, PDR is a major cause of blindness in adults and is also caused by the growth of abnormal blood vessels. Importantly, the Phase I Study found that OC-10X can be safely applied topically in human eyes without adverse ocular or systemic effects.

Currently, there are few options for the treatment of PDR. Clinical options, such as laser photocoagulation or vitrectomy, require surgery and can permanently impair patients' vision. With few treatment options available, administration of OC-10X as a topical therapy, along with its novel mechanism, has the potential to provide benefits to patients with ocular diseases associated with angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients diagnosed with Proliferative Diabetic Retinopathy will be eligible if the following inclusion criteria are met:

1. Ability to provide approved written informed consent and complies with study-related procedures/assessments for the full duration of the study, having age ≥18 years.
2. Type 1 or Type 2 Diabetes Mellitus.
3. Proliferative Diabetic Retinopathy (level 61, 65, 71, or 75) in one or both eyes without evidence of significant vitreous/pre retinal hemorrhage that would limit photographic documentation of area of neovascularization and without pre-retinal fibrosis. If both eyes meet eligibility requirements, the less affected eye will be selected to receive investigational drug or placebo. The second eye will be treated with the standard of care. (e.g. panretinal laser photocoagulation).
4. Best-Corrected Visual acuity of 20/200 or better in each eye.
5. If female and:

   * Of childbearing potential, agrees to use an acceptable method of birth control as judged by the Investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), for the duration of the study and for at least 2 weeks following the final dose of study drug or abstinence; or
   * Is postmenopausal for at least 1 year; or
   * Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
   * Is not pregnant or breastfeeding.

Exclusion Criteria:

Male or female patients diagnosed with Proliferative Diabetic Retinopathy will not be eligible in the study if any of the exclusion criteria are met:

1. Clinically significant systemic diseases/conditions that, in the opinion of the Investigator, could negatively affect the safety of the patient during the study on a as determined on a case by case basis (e.g., unstable medical status including uncontrolled blood pressure, cardiovascular disease, uncontrolled liver disease, glycemic control or significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant, hepatic, pulmonary, gastrointestinal or neurological diseases, cancer or BMI).
2. Participation in any other clinical study/trial within the past 30 days prior to randomization.
3. Current treatment for active systemic infection.
4. Known allergy to any component of the formulation or to topical anesthetics (e.g., benzalkonium chloride, fluorescein, etc.).
5. History of any psychiatric illness, which may impair the ability to provide written informed consent.
6. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
7. Positive for urinary screen testing of drugs of abuse (opiates, cannabinoids, amphetamines, barbiturates, benzodiazepines, cocaine).
8. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
9. Use of anti-mitotic or anti-metabolite therapy within 2 months of enrollment.
10. Planned use of any ocular or systemic medications that the Investigator determines unacceptable during the study (i.e. anti-vascular endothelial growth factor [VEGF] therapy), with the exception of oral contraceptives and short-term use of over-the-counter analgesics during the study.
11. Any other concurrent condition that, in the opinion of the Investigator, would prevent completion of the clinical trial, including inability to comply with the study requirements.
12. Presence of significant fibrosis or gliosis of the neovascularization of the disc or retina.
13. Presence of tractional retinal detachment.
14. History of panretinal laser photocoagulation (PRP) for Proliferative Diabetic Retinopathy.
15. Patients likely to require treatment for diabetic macular edema during the study.
16. Any intraocular surgery or trauma within 6 months before trial enrollment.
17. History of chronic ocular disease that, in the opinion of the Investigator, will affect neovascular progression.
18. Myocardial infarction, other cardiac events requiring hospitalization, stroke, transient ischemic attack, or treatment for congestive heart failure within 6 months prior to randomization that, in the in the opinion of the Investigator, could negatively affect the safety of the patient during the study.
19. Current use of contact lenses.
20. Concurrent or anticipated use of ocular agents during the study period that are considered by the Investigator to interfere with the study objectives.
21. History or evidence of ocular infection, inflammation, blepharitis, or conjunctivitis within 2 months; history of herpes simplex keratitis.
22. An ocular condition is present (other than diabetes) that, in the opinion of the Investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
23. Substantial cataract that,

    * In the opinion of the Investigator, is likely to be causing decreased visual acuity by 3 lines or more (e.g.., cataract reducing acuity to 20/40 or worse).
    * Would interfere with photography of the retina.
24. Aphakia, uncontrolled glaucoma (in Investigator's judgment).
25. Inability to tolerate eye drops in the eye or to have eye drops correctly administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by the mean change of area of neovascularization of the disc (NVD) from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by the mean change of area of neovascularization of the disc (NVD) from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by the change of area of neovascularization elsewhere in the retina (NVE) from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by the change of area of neovascularization elsewhere in the retina (NVE) from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by the change of area of "Posterior NVE" from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by the change of area change of area of "Posterior NVE" from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by regression of total area of neovascularization (NVD+NVE) from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  The effect of OC-10X 2% on regression/inhibition of neovascularization in PDR patients as measured by regression of total area of neovascularization (NVD+NVE) from baseline compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.

SECONDARY OUTCOMES:
Change from baseline of regression of intraretinal microvascular abnormalities (IRMA) in PDR patients as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of intraretinal microvascular abnormalities (IRMA) in PDR patients as compared to Visit 6 (Week 24)for OC-10X 2% vs. Placebo.
Change from baseline of regression of intraretinal hemorrhage as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of intraretinal hemorrhage as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of regression of venous beading as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of venous beading as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of regression of area of capillary non-perfusion beading as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of area of capillary non-perfusion beading as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of regression of intraretinal exudation (lipid) as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of intraretinal exudation (lipid) as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of regression of macular edema (central subfield thickness) as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of macular edema (central subfield thickness) as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of regression of macular volume as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of regression of macular volume as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of best-corrected ETDRS visual acuity as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of best-corrected ETDRS visual acuity as compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Change from baseline of macular thickness as measured by Optical Coherence Tomography (OCT) compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo. | Baseline - 24 weeks
  Change from baseline of macular thickness as measured by Optical Coherence Tomography (OCT) compared to Visit 6 (Week 24) for OC-10X 2% vs. Placebo.
Number of patients requiring rescue treatment at the end of the study. | Baseline - 24 weeks
  Number of patients requiring rescue treatment at the end of the study.
Number of patients requiring pars plana vitrectomy surgery due to presence of vitreous hemorrhage at the end of the study. | Baseline - 24 weeks
  Number of patients requiring pars plana vitrectomy surgery due to presence of vitreous hemorrhage at the end of the study.
Number of patients requiring pars plana vitrectomy surgery due to traction retinal detachment at the end of the study. | Baseline - 24 weeks
  Number of patients requiring pars plana vitrectomy surgery due to traction retinal detachment at the end of the study.

OTHER OUTCOMES:
Change from baseline of how the eye feels as assessed by patient query. | Baseline - 24 weeks
  Change from baseline of how the eye feels as assessed by patient query.
Change from baseline of evaluation of corneal epithelium, bulbar and lower conjunctiva by biomicroscopy. | Baseline - 24 weeks
  Change from baseline of evaluation of corneal epithelium, bulbar and lower conjunctiva by biomicroscopy.
Change from baseline of evaluation of vital signs (body temperature, pulse rate blood pressure and respiratory rate). | Baseline - 24 weeks
  Change from baseline of evaluation of vital signs (body temperature, pulse rate blood pressure and respiratory rate).
Evaluation of systemic exposure as measured by bioanalytic methods. | Baseline - 24 weeks
  Evaluation of systemic exposure as measured by bioanalytic methods.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia B Williams, PhD, Study Director — OcuCure Therapeutics, Inc.
Locations (1):
- Bangladesh Eye Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided